CLINICAL TRIAL: NCT02401451
Title: SL-AF Trial - (Six Lead Identification of Atrial Fibrillation [AF])
Acronym: SL-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiocity Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ACB1-1001-1941; NCT02124629 (obsolete NCT alias)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ECG acquisition (Experimental): ECG acquisition using the standard ECG machine
  Intervention: An ECG will be performed on every participant using the novel device called the 'RhythmPadGP'
  Interventions: Device: RhythmPadGP

INTERVENTIONS:
Device: RhythmPadGP — ECG acquisition using a novel device RhythmPadGP

SUMMARY:
The 12-lead ECG is an essential tool in cardiovascular assessment. Novel technology has the potential to improve the diagnostic yield of arrhythmias, whilst improving the patient experience.

The RhythmPadGP is a novel device which acquires a 6-lead ECG without the need for the patient to undress.

The aim of the study is to assess the ability of the device to diagnose cardiac rhythms.

Simultaneous recording of the RhythmPadGP 6-lead ECG will be undertaken at the same time as the standard 12-lead ECG.

The 12-lead ECGs and 6-lead ECGs will be analysed by a Cardiologist, who will be blinded to each set of ECGs and the automated diagnostic report produced by the RhythmPadGP device.

Such a novel diagnostic tool could replace the standard 12-lead ECG for rapid assessment and diagnosis of arrhythmias. Additionally, as calls for a national screening programme to detect atrial fibrillation (and prevent AF-related thromboembolism) currently intensify, the RhythmPad has the potential to revolutionise how we screen our patients.

DETAILED DESCRIPTION:
The concept for the Rhythm Pad is to screen the public non-invasively for a cardiac rhythm abnormality, every time that they interact with a clinician. Cardiocity have conducted significant trialing of the RhythmPad product within both the primary care setting at the Old Cottage Hospital in Epsom and in a secondary care setting at St Peter's Hospital in Chertsey. The initial results were encouraging with a simple hand screening providing an indication of AF in 66% of the confirmed cases of AF, when verified by a traditional electrocardiogram (ECG) known as a GE MAC550 12 lead device as the benchmark.

The main aim is for the RhythmPad range of products to increase the ability to diagnose cardiac rhythm abnormalities, along with reducing the number of false positive referrals to secondary care for a 12 lead Electrocardiogram of ECG. As such confirming the diagnosis before referral reduces the number of false positive referrals. If one of our algorithms thinks that there is evidence that the person might be in a state of Atrial Fibrillation (AF), Flutter, might have left or right bundle branch block, etc, then by moving to the 6 lead we are able to increase the confidence of the diagnosis.

The RhythmPad is now able to support a 6 lead ECG acquisition, this is by using a modified device called the RhythmPadGP as such we would plan to trial this technology with St Peter's Hospital. We have learnt from the experiences of the previous trails. We know that 5% of the entire population will not have strong enough Lead 1 ECG when measured from their hands. Also those with Essential Tremor, Parkinson's etc. are not able to keep their hands steady for an accurate reading to be taken. In such cases, or as an escalation from the one lead data, we now offer through a simple Velcro ankle strap attachment the ability to record 6 leads of data.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years of age
* able to consent
* attending to St Peter's Hospital for an ECG
* No known allergies to the velcro or metal used in the RhythmPadGP leads

Exclusion Criteria:

* Age less than 18 years of age
* Not able to consent
* Allergies to the metal/velcro strap
* Medical condition affecting the wrists that may be interfered with by the attachment of the RhythmPdGP leads, such as a fractured limb that has a cast
* Those with pacemakers or other implanted cardiac devices that would interfere with the ECG recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Six Lead Identification of Atrial Fibrillation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Riyaz A Kaba, MBBS, Principal Investigator — Ashford and St Peter's Hospitals NHS Foundation Trust
Locations (1):
- Ashford and St Peters NHS Trust, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided